CLINICAL TRIAL: NCT03180385
Title: Neurally Adjusted Ventilatory Assist (NAVA) Versus Conventional Biphasic Positive End Expiratory Pressure (BiPAP) Non-Invasive Respiratory Support in Infants Following Congenital Heart Surgery
Brief Title: NAVA Versus BiPAP Non-Invasive Respiratory Support in Infants Following Congenital Heart Surgery
Acronym: NAVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very small percentage of enrolled patients needing non-invasive support and small chance of us reaching target enrollment within funding period.
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1701-008
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2019-10-15 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Failure
Keywords: NAVA; BiPAP; Pediatrics; Cardiac Surgery
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Neurally-Adjusted Ventilatory Assist (NAVA) (Experimental): Synchronized biphasic non-invasive respiratory support
  Interventions: Device: Neurally-Adusted Ventilatory Assist (NAVA)
- Biphasic Positive Airway Pressure Support (BiPAP) (Active Comparator): Conventional non-invasive respiratory support
  Interventions: Device: Biphasic Positive Airway Pressure Support (BiPAP)

INTERVENTIONS:
Device: Neurally-Adusted Ventilatory Assist (NAVA) — Delivery of positive pressure is based on the electrical activity of the diaphragm (Edi) via a nasogastric (NG) catheter that is placed on the phrenic nerve, which runs along the esophagus. This results in synchronous ventilation for the patient.
  Arms: Neurally-Adjusted Ventilatory Assist (NAVA)
Device: Biphasic Positive Airway Pressure Support (BiPAP) — Conventional form of non-invasive respiratory support that does not deliver positive airway pressure in a synchronous fashion.
  Arms: Biphasic Positive Airway Pressure Support (BiPAP)

SUMMARY:
Pediatric patients often require prolonged mechanical ventilation after cardiac surgery which comes with many undesirable effects. As a result, neurally-adjusted ventilatory assist (NAVA) and biphasic positive airway pressure support (BiPAP) have been developed as non-invasive alternatives to providing respiratory support post-operatively. The investigators hypothesize that providing synchronized biphasic support with NAVA will be associated with shorter duration of non-invasive respiratory support, less sedation requirements, and reduced length of hospital stay. This is a prospective, randomized study. Subjects are randomized to receive either NAVA or BiPAP following their cardiothoracic surgery.

DETAILED DESCRIPTION:
Mechanical ventilation is often very necessary in the care of critically ill pediatric patients. However, it comes with many different complications that include chronic lung disease, tissue damage, and ventilator-associated pneumonia. Over time, we have increased our understanding of how a child's physiology interacts with a ventilator and this has led to two different non-invasive forms of respiratory support: bilevel positive air pressure (BiPAP) and neurally adjusted ventilator assist (NAVA). While both modalities come with a lot of benefits such as improved gas exchange, decreased respiratory and heart rate and decreased inspiratory work of breathing, NAVA has the ability to provide synchronous ventilatory support due to the electrical activity of the diaphragm.

The purpose of this study is to compare clinical outcomes following use of NAVA versus BiPAP in patients undergoing cardiac surgery, Specifically, comparisons of non-invasive respiratory support, duration of sedation, and length of hospital stay. The investigators hypothesize that the use of NAVA will lead to a shorter duration of non-invasive respiratory support, less sedation requirements, and reduced length of hospital stay compared to the use of BiPAP.

This is a single-site, prospective randomized study. Subjects are randomized into two arms: those who receive NAVA and those who receive BiPAP post-operatively.

Subjects will be followed for up to 14 days post-operatively or until they are discharged, whichever comes first. Pain medication administered, FLACC (Face, Legs, Activity, Cry, Consolability), and SBS (State Behavioral Scale) scores are recorded daily for up to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative cardiac surgery patients admitted to the Cardiovascular Care Center (CVCC) at Children's Hospitals and Clinics of Minnesota
* Recommended for non-invasive (NIV) respiratory support following extubation, per provider discretion
* 0 to 12 months of age

Exclusion Criteria:

* Documented airway malformation (congenital or acquired)

  1. Laryngomalacia
  2. Bronchomalacia
  3. Laryngeal web
  4. Tracheal or bronchial rings (complete or incomplete)
* Documented ENT abnormality
* Documented central apnea
* Patients who are overly sedated, per provider discretion
* Tracheostomy in place at time of cardiac surgery
* Documented phrenic nerve paralysis (Note: Vocal cord paresis and paralysis will not be an exclusion)
* Other chromosomal abnormality (non-Down syndrome)
* Chronic lung disease
* Pre-operative non-invasive respiratory support

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen A McGuire, RN, MSN, CPNP-AC, Principal Investigator — Children's Hospitals and Clinics of Minnesota; Robert Horvath-Csongradi, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed consent was obtained for 15 participants. However, the reason there are only 2 participants listed under "total started in participant flow" is because these were the only participants who were actually randomized. The other 13 participants were extubated and did not need BiPAP/NAVA. They were not randomized and were excluded.
Period: Overall Study
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients who were enrolled in the study and needed non-invasive respiratory support post-cardiac surgery were randomized to NAVA, only BiPAP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP) | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 0.46 (0.04) | 0.46 (0.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Average Post-operative Midazolam Dose
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
mg/kg |  | 0.035 (0.007)

2. Primary Outcome: Post-operative Pain Scores-FLACC
Description: FLACC (Face, Legs, Activity, Cry, Consolability) scale
Time Frame: Up to 14 days post-operatively
Population: There were no FLACC scores in the electronic medical record for either of these 2 participants so this is why there are no results reported.
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Post-operative Sedation Scores-SBS
Description: SBS (State Behavioral Scale)
Time Frame: Up to 14 days post-operatively
Population: There were no SBS scores in the electronic medical record for either of these 2 participants so this is why results were not reported.
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Length of Intubation
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
hours |  | 37.24 (3.87)

5. Primary Outcome: Length of Non-Invasive Respiratory Support
Time Frame: Up to 14 days post-operatively
Population: For this outcome, data for only one participant is available
Measure: Number; unit: hours
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 1
hours |  | 7.17

6. Primary Outcome: Average Post-operative Morphine Dose
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
mg/kg |  | NA (NA) — Both participants did not receive morphine for pain control

7. Primary Outcome: Average Post-operative Lorazepam Dose
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
mg/kg |  | 0.11 (0.15)

8. Primary Outcome: Average Post-operative Dexmedetomidine Dose
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
mcg/kg |  | 6.71 (9.49)

9. Primary Outcome: Average Post-operative Total Fentanyl Dose
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
mcg/kg |  | 8.09 (7.06)

10. Primary Outcome: Average Post-operative PCA Fentanyl Dose
Time Frame: Up to 14 days post-operatively
Population: All patients who were randomized ended up in the BiPAP group and not the NAVA group.
Measure: Mean (Standard Deviation); unit: boluses
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
Number analyzed (Participants) | 0 | 2
boluses |  | NA (NA) — Both participants did not receive PCA boluses of fentanyl for pain control

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the span of the patient's hospital stay, specifically up to 14 days post-cardiac surgery.
Description: Adverse events were assessed via review of daily progress notes by both cardiology and cardiac intensive care providers within the electronic medical record (EMR).
Arm/Group | Neurally-Adjusted Ventilatory Assist (NAVA) | Biphasic Positive Airway Pressure Support (BiPAP)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurally-Adjusted Ventilatory Assist (NAVA) (N=0) | Biphasic Positive Airway Pressure Support (BiPAP) (N=2)
Re-intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient had desaturation episode to 29% and was subsequently re-intubated on post-operative day #2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT03180385/Prot_SAP_000.pdf